CLINICAL TRIAL: NCT02572115
Title: Differentiated Access to Out-of-hours Primary Care Through Emergency Access
Acronym: Akutknappen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); Emergency Medical Services, Capital Region, Denmark (Other Government); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JFME001
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-09

CONDITIONS: After-hours Care
Keywords: After-Hours Care; Primary Care; Emergency Medical Services/utilization; Denmark; Questionnaires; Patient Satisfaction; Patient feeling of safety; Triage/standards; Referral and Consultation/statistics & numerical data; Humans; Male; Female; Hotlines; telenursing; Night Care/utilization; postal service
MeSH Terms: conditions — Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm - jumped the line (Active Comparator): This arm is presented with the possibility to use the "emergency access button" that enables the patient to bypass the telephone waiting line. This arm represents the patients who choose to use the intervention.
  Interventions: Behavioral: Akutknappen - used
- Intervention arm - did not jump the line (Active Comparator): This arm is presented with the possibility to use the "emergency access button" that enables the patient to bypass the telephone waiting line. This arm represents the patients who got the option to use the intervention but DID NOT.
  Interventions: Behavioral: Akutknappen - not used
- Control (No Intervention): This arm does not get the intervention.

INTERVENTIONS:
Behavioral: Akutknappen - used — A caller chooses to bypass the telephone waiting line by pressing the emergency access button
  Arms: Intervention arm - jumped the line
Behavioral: Akutknappen - not used — A caller chooses NOT to bypass the telephone waiting line.
  Arms: Intervention arm - did not jump the line

SUMMARY:
The purpose of this randomized controlled trial is to test the use of an emergency button that allows patients to jump the telephone waiting line at the out-of-hours primary care in two regions in Denmark if they perceive their illness as acute and severe.

DETAILED DESCRIPTION:
Patients calling the Danish out-of-hours primary care service (OOH-PC; i.e. lægevagt) and Medical Helpline 1813 (i.e. Akuttelefonen) queue up in the telephone waiting line. Ranging from patients calling for acute illness such as chest pain to parents calling to ask if their coughing child is well enough to go to day care the next day, they must all wait for their turn to talk to the triage general practitioner (GP) or triage nurse. This Project is a part of a PhD-project which is a composition of two different randomised controlled studies with overlapping background. This registration with www.clinicaltrials.gov only concerns the following study:

- Intervention to bypass the telephone queue in case of a perceived emergency: The investigators implement an option for patients to bypass the telephone queue by pressing a button if they perceive their illness as acute and severe.

Background:

Acute out-of-hours (OOH) care is an important part of health care and the point of entrance into the health care system for many patients, who contact outside normal working hours (i.e. 4 pm to 8 am on weekdays, all weekends, and bank holidays). Patients with acute health problems have several options to access the health care system, such as OOH-PC, 112-Emergency Medical Communication Centre (112-EMCC), and Medical Helpline 1813. These settings have complementary aims in delivering health care, but at the same time their patient population is partly overlapping.

Primary care is often the first point of contact, also outside office hours. However, in the Capital Region of Denmark patients call the Helpline 1813 which is answered by triage nurses who have the option to forward the call to a doctor, to triage to a consultation at the emergency department (ED) or another hospital department, to order a home visit, to forward the call to 112-EMCC or to give telephone health advice. In the four other regions OOH-PC is run by GPs, who answer and triage all telephone calls. They can triage to a telephone advice, a clinic consultation, a home visit, or directly refer to the ED/hospital. Patients contacting the OOH-PC or Helpline 1813 are put on hold and wait in a telephone queue if no GP or nurse is available to answer their call.

The Danish acute care settings are intended to provide care to different patient groups depending upon the nature and severity of the health problem. With the decision to contact a specific setting, patients themselves choose the point of access to acute care, thus influencing their care pathway. An 'inappropriate´ choice may result in serious delay of treatment or insufficient intensive care, if they for example contact primary care instead of 112-EMCC in life-threatening cases. On the contrary, over-use or -treatment is a potential risk if calling 112-EMCC for minor problems.

At the moment, if a patient calls OOH-PC or Helpline 1813, he has to wait in line, even if the health problem is experienced as highly urgent or life-threatening. The alternative to waiting in line is calling 112-EMCC instead, as there is no possibility to bypass the telephone waiting line. In the Netherlands this functionality is integrated in the telephone system, meaning that patients who jump the waiting line are connected to the first available telephone triage professional.

No information is available about the number of patients whose safety has been compromised because of extensive waiting. The investigators also lack knowledge on the number of patients who decide to contact another health care service, such as 112-EMCC, due to the waiting time in OOH-PC and Helpline 1813. At the OOH-PC about 5% of patients estimate their condition as potentially life-threatening and approximately 1% of all telephone contacts are directly triaged to 112-EMCC. In the Central Denmark Region this accounts for approximately 7,000 patient contacts per year who may experience potential harm from a delay as a consequence of the telephone queue.

Although it is not clear whether the absence of the possibility to jump the line is a problem for patients, its presence may provide patients with a feeling of safety and reduce the level of stress in medical situations which are experienced as distressing.

Aim:

To implement the jump-the-line option in OOH-PC and Medical Helpline 1813 to:

1. study the frequencies of patients jumping the line and the general characteristics of these patients,
2. study the patients' reasons for jumping the line and their satisfaction with this option,
3. evaluate the amount of jumps assessed as relevant by the triage GP/nurse

Methods

Design, setting and intervention:

The investigators conduct a randomised controlled trial (RCT) at OOH-PC in the Central Denmark Region and Helpline 1813 in the Capital Region. The two settings are used so the investigators can make a comparison of the usage of the jump-option in the two regions and hopefully a well-founded recommendation regarding the intervention. At the moment, when calling, patients are already routinely asked to press their CPR number at the telephone. Hereafter, the patients will be randomized into two arms according to their date of birth (even or uneven date in the month) which is part of the Social security number (Central Person Register, CPR number).

For those in the intervention arm, the message at the answering machine will inform the patient of the possibility to jump the waiting line by pressing '9'. By doing this their call will be answered by the next available triage person. On the computer screen of the triage person a message will appear, if the patient has used the jump option. Patients at the control arm will get the normal message at the answering machine and will not get the possibility to jump the line. If patients call several times during the study period they will be randomized to the same arm every time, using the CPR number. If patients do not press their CPR number, they will get the normal message at the answering machine without the option to jump the line.

Data collection:

A questionnaire will pop-up on the PC for the triage GPs in the Central Region of Denmark and triage nurses and doctors in the Capital Region for all patients who use the jump option. This pop-up questionnaire contains questions about the medical and social relevance of jumping the line, the degree of urgency, the reason for encounter (RFE) and the probable diagnosis. The questionnaire is short and can be completed in less than a minute. Furthermore, a similar questionnaire (without the question about the relevance for jumping the line) will pop-up for the triage professionals for a random group of patients in the intervention arm who did not jump the line and for a random group of patients belonging to the control arm. This will enable the investigators to compare the three groups. This method of collecting data from the GPs has been found feasible in earlier studies.

A patient questionnaire will be sent to a random group of patients who use the jump option. Questions focus on the reason for using the jump option, patient satisfaction, and the effect of the intervention on their feeling of safety, as well as relevant patient and contact characteristics (e.g. RFE). Furthermore, questionnaires will be sent to a random group of patients from the intervention arm who did not jump the line. Questions for this group focus on the reason for not using the jump option, RFE, patient satisfaction, and the effect of the intervention on their feeling of safety. Finally, a questionnaire will be sent to a random group of patients in the control group, focusing on the RFE and patient satisfaction with the current system.

As a part of the telephone message in the OOH-PC telephone, patients will be informed about the ongoing study with the option not to participate in the study. The questionnaires are planned to be sent in a few days after the contact by ordinary letter as well as by a message to the patient's electronic mailbox required by the state (e-boks) with a link to an electronic version of the questionnaire. If the patient is less than 14 years old, the questionnaire will be addressed to the parents. Patients will only receive one questionnaire in the study period although they may have several contacts.

Furthermore, the investigators collect information of all contacts to OOH-PC and Helpline 1813 in the study period the electronic patient record system of OOH-PC and Helpline 1813 can provide: CPR number of the patient, date and time of contact, triage outcome (i.e. telephone consultation, consultation, home visit or referral to ED or other hospital departments), use of jump the line option, and waiting time in the telephone line at time of patient call to the service. If the patient has chosen to jump the line, the investigators also collect the length of waiting time at the time of the jump.

Study period and power calculation:

Based on the patient questionnaires: The investigators want to be able to detect a minimum mean difference of 0.3 between jumpers and non-jumpers in the outcome measures regarding satisfaction and feeling of safety. If the investigators assume that the sample standard deviation is 1, significance level is 5%, power is 95% and given a mean of 3 the investigators need a total of 580 answered patient questionnaires to be able to detect a difference of 0.3 between the two groups. This means that, with a response rate from the patients of 40%, the investigators have to send out 1450 questionnaires.

In 2013 the total number of contacts with OOH-PC in the Central Denmark Region was approximately 660,000. An earlier study showed that approximately 80% of patients type in their CPR number on their phone when calling the service. Numbers from the Netherlands show a user rate of 3 % of their version of the option to jump the line. An estimated response rate from the GPs of 70% gives a study period of approximately 1,6 months.

Based on number of jumps: In relation to the aim of frequency of jumping the line the investigators want to determine the user rate. The investigators estimate a user rate of 3 % and this gives them 7,800 users of the intervention in one year. In order to obtain satisfactory power in the calculations of the usage of the jump option the investigators want a 95%-confidence interval of +/- 2,2%. This means that the investigators need at least 1950 jumpers, which requires 3 months to complete the study.

In conclusion the investigators need approximately 3 months to complete the study if they want satisfactory power regarding the frequency of jumps and patient satisfaction.

The investigators plan to conduct a pilot study with a running time of 1-2 weeks to give a more precise estimate of the user rate in order to perform a more accurate power calculation to define the length of the study period.

Analyses:

The investigators provide a descriptive analysis of the group of patients who jump the line, the group who chose not to jump the line, and patients from the control group, along with univariate analyses comparing the patients in the three groups (i.e. patient characteristics, RFE, incentives). Descriptive analyses will be performed using Student's t-test for data following a normal distribution, Mann-Whitney U-test for non-normally distributed data, and chi-square test for categorical data. For the primary outcome measures patient satisfaction and feeling of safety the investigators perform intention to treat analyses as wells as analyses between subgroups. The association between relevant jumps and GP assessed level of urgency and patient characteristics is explored by the use of multivariate binomial regression taking clustering at GP level into account. The association between patients' choosing to jump the line, satisfaction with having the option, and the reasons to do so, is assessed using multivariate binomial regression models.

Perspective:

This study will provide knowledge on the feasibility and effects of implementing an option to jump the telephone waiting line at OOH-PC and Helpline 1813, and it will be clarified whether patients will use such an option appropriately. This information will be used to decide whether this intervention should be implemented nationwide. The percentage of patients potentially benefiting from this option to jump the line is expected to be relatively limited, but as the total number of contacts with OOH-PC is extensive, the absolute number of patients actually benefiting from this simple intervention is likely to be substantial. Especially in the area of feeling safety the investigators hope to see a significant effect.

This intervention is robust and can be extended to other regions and settings easily. Information about the decrease in waiting time for urgent cases could lead to stratification of quality goals for different patient groups. Also a higher number of cases with acute illness could be handled by the OOH-PC which could ease the pressure on 112-EMCC.

ELIGIBILITY:
Inclusion Criteria:

* All patients calling the OOH-PC in the Central Region of Denmark and the Helpline 1813 in the Capital Region in the study period are included

Exclusion Criteria:

* patients who died
* patients from 14 to 17 years (they sometime contact the services without the knowledge of their parents and receiving a questionnaire at their home address could be inconvenient)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7385 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction and feeling of safety with the intervention measured by questionnaire | Measured by questionnaire after contact with the OOH-PC sent out 2-4 days after contact
Frequencies of patients who jumped the line | Up to 4 months
  Numbers and statistics from data provider

SECONDARY OUTCOMES:
Description of the characteristics of the patients who jump the line compared with the ones who do not | Measured by questionnaire after contact with the OOH-PC sent out 2-4 days after contact
  The patients answer a questionnaire with info about age, gender, reason for encounter, ethnicity, education etc. This is to give a general description of the ones who use the intervention. It is not possible to single out every variable as an individual outcome measure.
Reasons for jumping (or not jumping) the line measured by questionnaire | Measured by questionnaire after contact with the OOH-PC sent out 2-4 days after contact
  Above mentioned questionnaire contains questions about reasons for jumping the line
Rate of jumps assessed as relevant by the triage professional | Up to 4 months
  Triage GPs and nurses answer pop-up questionnaires on their workstation after each contact.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Christensen, MD, PhD, Study Director — Section for General Practice, University of Aarhus; Morten B Christensen, MD, PhD, Study Chair — Research Unit for General Practice, University of Aarhus; Linda Huibers, MD, PhD, Study Chair — Research Unit for General Practice, University of Aarhus; Freddy Lippert, MD, Study Chair — Prehospital Unit, Capital Region of Denmark
Locations (1):
- Research unit for General Practice, University of Aarhus, Aarhus, Danmark, Denmark

REFERENCES:
- [Background] Flarup L, Moth G, Christensen MB, Vestergaard M, Olesen F, Vedsted P. A feasible method to study the Danish out-of-hours primary care service. Dan Med J. 2014 May;61(5):A4847. PMID 24814746
- [Background] Christensen MB, Skafte-Holm P, Weinicke HH, Greibe J, Rem J, Sauer M, Andersen DH, Gliese MS. [General practitioners' evaluation of the out-of-hours service in Copenhagen County]. Ugeskr Laeger. 2005 Sep 5;167(36):3412-5. Danish. PMID 16159495
- [Background] Christensen MB, Olesen F. Out of hours service in Denmark: evaluation five years after reform. BMJ. 1998 May 16;316(7143):1502-5. doi: 10.1136/bmj.316.7143.1502. PMID 9582141
- [Background] Bunn F, Byrne G, Kendall S. Telephone consultation and triage: effects on health care use and patient satisfaction. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD004180. doi: 10.1002/14651858.CD004180.pub2. PMID 15495083
- [Background] Giesen P, Smits M, Huibers L, Grol R, Wensing M. Quality of after-hours primary care in the Netherlands: a narrative review. Ann Intern Med. 2011 Jul 19;155(2):108-13. doi: 10.7326/0003-4819-155-2-201107190-00006. PMID 21768584
- [Background] Huibers L, Koetsenruijter J, Grol R, Giesen P, Wensing M. Follow-up after telephone consultations at out-of-hours primary care. J Am Board Fam Med. 2013 Jul-Aug;26(4):373-9. doi: 10.3122/jabfm.2013.04.120185. PMID 23833151
- [Background] Huibers L, Moth G, Andersen M, van Grunsven P, Giesen P, Christensen MB, Olesen F. Consumption in out-of-hours health care: Danes double Dutch? Scand J Prim Health Care. 2014 Mar;32(1):44-50. doi: 10.3109/02813432.2014.898974. PMID 24635578
- [Background] Huibers L, Thijssen W, Koetsenruijter J, Giesen P, Grol R, Wensing M. GP cooperative and emergency department: an exploration of patient flows. J Eval Clin Pract. 2013 Apr;19(2):243-9. doi: 10.1111/j.1365-2753.2011.01806.x. Epub 2012 Feb 5. PMID 22304568
- [Background] Murphy AW. 'Inappropriate' attenders at accident and emergency departments I: definition, incidence and reasons for attendance. Fam Pract. 1998 Feb;15(1):23-32. doi: 10.1093/fampra/15.1.23. PMID 9527294
- [Derived] Ebert JF, Huibers L, Christensen B, Collatz Christensen H, Christensen MB. Does an emergency access button increase the patients' satisfaction and feeling of safety with the out-of-hours health services? A randomised controlled trial in Denmark. BMJ Open. 2020 Sep 30;10(9):e030267. doi: 10.1136/bmjopen-2019-030267. PMID 32998912
- [Derived] Ebert JF, Huibers L, Christensen B, Lippert FK, Christensen MB. Do callers to out-of-hours care misuse an option to jump the phone queue? Scand J Prim Health Care. 2019 Jun;37(2):207-217. doi: 10.1080/02813432.2019.1608067. Epub 2019 May 9. PMID 31070507
- [Derived] Ebert JF, Huibers L, Lippert FK, Christensen B, Christensen MB. Development and evaluation of an "emergency access button" in Danish out-of-hours primary care: a study protocol of a randomized controlled trial. BMC Health Serv Res. 2017 May 31;17(1):379. doi: 10.1186/s12913-017-2308-y. PMID 28566087
- See also: Danish statistics — http://statistikbanken.dk